CLINICAL TRIAL: NCT04933669
Title: Prospective Multicenter Clinical Study of Neoadjuvant Imatinib Mesylate for Gastrointestinal Stromal Tumors
Acronym: ZJGIST-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Yu jiren, Chief of Gastrointestinal Surgery, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210023C-R1
Record Dates: First submitted 2021-06-09; First posted 2021-06-22 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Progression-free Survival; Gastrointestinal Stromal Tumor; Neoadjuvant
Keywords: Progression-free survival; Gastrointestinal Stromal Tumors; neoadjuvant
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imatinib neoadjuvant (Experimental): Patients receive oral imatinib mesylate 400mg once daily for 3-12 months in the absence of disease progression or unacceptable toxicity. Within 1 week after completion of preoperative imatinib mesylate, patients with responding or stable disease undergo surgical resection. After complete resection, patients receive oral imatinib mesylate 400mg once daily for 36 months in the absence of disease progression or unacceptable toxicity, and are followed for 5 years.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib neoadjuvant therapy
  Other Names: neoadjuvant therapy

SUMMARY:
The R0 resection rate of gastrointestinal stromal tumor (GIST) with high recurrence risk was relatively low, and the relapse-free survival rate was relatively low, which needed to be further improved. A few retrospective analyses and a small sample of prospective studies have found that neoadjuvant therapy with imatinib mesylate can improve R0 resection rates. Whether neoadjuvant therapy prolongs long-term survival remains unclear. The primary objective of this study was to evaluate 5-year progression-free survival (PFS) for GIST patients with high recurrence risk after neoadjuvant treatment with imatinib mesylate.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative histologically confirmed primary gastrointestinal stromal tumor
* Tumor must stain positive for c-Kit (CD117) and/or discovered on gist-1 (DOG-1) by immunohistochemistry
* Gene mutation test report including c-kit exons 9,11,13 and 17 and platelet-derived growth factor receptor alpha (PDGFRA) exons 12 and 18
* High risk GIST (as modified National Institutes of Health (NIH) 2008): stomach (maximum tumor diameter> 10.0cm), nonstomach (maximum tumor diameter> 5.0cm)
* Gender is not limited. Age: ≥ 18 years and ≤ 80 years old
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-1
* Patient had informed consent and signed a written consent form

Exclusion Criteria:

* Asp842Val (D842V) mutation in Exon 18 of PDGFRA gene, or wild type (c-kit exon 9,11,13,17, and PDGFRA Exon 12,18), or c-kit exon 9 mutation
* Treated with tyrosine kinase inhibitors including Imatinib
* Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT)>2.5×ULN(upper limit of normal)，or Total bilirubin (TBIL)>1.5×ULN，or Creatinine (Cr)>1.0×ULN
* Absolute neutrophil count (ANC) < 1.5 × 10 ^ 9 / L；or Platelet count (PLT) < 75 × 10 ^ 9 / L；or Hemoglobin (Hb) ≥ 90 g / L
* Previous or concurrent other active malignant tumors (except for basal cell carcinoma of the skin, or cervical cancer in situ that has undergone curative therapy)
* Distant metastases are present
* Any of the following conditions during the 12 months prior to entry: myocardial infarction, severe / unstable angina, coronary artery / peripheral artery bypass surgery, symptomatic congestive heart failure, or cerebrovascular accidents
* positive Human Immunodeficiency Virus (HIV) antibody
* Currently participating in other clinical trials
* Pregnant or lactating women or have fertility without taking contraception
* Suffering from other serious acute and chronic physical or mental problems, or abnormal laboratory tests, will increase the risk of participation or drug use, or interfere with the judgment of the findings, judged by the researchers as participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival（PFS） | 5 years
  Progression free survival（PFS）

SECONDARY OUTCOMES:
Overall survival（OS） | 5 years
  Overall survival（OS）
Objective Response Rate （ORR） | Up to 1 year
  Rate of complete and partial response according to Choi criteria
R0 resection rate | Up to 1 year
  complete resection rate with microscopically negative margin

CONTACTS AND LOCATIONS:
Overall Officials: Jiren Yu, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No